CLINICAL TRIAL: NCT02734173
Title: Pilot Evaluation of the Influence of ABT450r, Ombitasvir, Dasabuvir +/- Ribavirin HCV Therapy on Insulin Resistance and Lipid Profile
Brief Title: Pilot HCV Direct Acting Antiviral Therapy and Metabolism
Acronym: 3D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20150305-01H
Record Dates: First submitted 2015-10-21; First posted 2016-04-12 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — ombitasvir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Genotype 1a Non-Cirrhotic Arm (Active Comparator): • 8 non-cirrhotic genotype 1a-infected recipients will receive a 12 week course of ABT450r-ABT267-ABT333 therapy plus ribavirin
  Interventions: Drug: ABT450r-ABT267-ABT333 +/- Ribavirin
- Genotype 1b Non-Cirrhotic Arm (Active Comparator): • 8 non-cirrhotic genotype 1b-infected recipients will receive a 12 week course of ABT450r-ABT267-ABT333 therapy without ribavirin
  Interventions: Drug: ABT450r-ABT267-ABT333 +/- Ribavirin
- Genotype 1a/1b Compensated Cirrhotic Arm (Active Comparator): • 8 compensated cirrhotic genotype 1a or 1b-infected recipients will receive a 12 week course of ABT450r-ABT267-ABT333 therapy plus ribavirin
  Interventions: Drug: ABT450r-ABT267-ABT333 +/- Ribavirin

INTERVENTIONS:
Drug: ABT450r-ABT267-ABT333 +/- Ribavirin — 12 week duration of HCV antiviral therapy with ABT450r-ABT267-ABT333 +/- Ribavirin
  Other Names: ombitasvir/paritaprevir/ritonavir, dasabuvir, ribavirin

SUMMARY:
There is compelling data supporting the pursuit of research into the effects of HCV antivirals on metabolic homeostasis. As a further rationale and justification, the experience with HIV antiretrovirals has clearly demonstrated that antiviral medications can produce profound changes in glucose metabolism, lipid profile and other measures of metabolic homeostasis. This establishes biological plausibility for this focus of research in HCV.

The new knowledge created from this research will:

1. Provide new information on the metabolic effects of the Abbvie 3D HCV antiviral regimen.
2. Provide insight as to whether there are metabolic advantages with RBV-free compared to RBV-containing HCV regimens. This is particularly relevant given the current uncertainty regarding the need for RBV in IFN-free, oral DAA regimens.
3. Provide insight into the impact of cirrhosis on metabolic milieu before, during and after HCV antiviral therapy

DETAILED DESCRIPTION:
There is a heavy burden of metabolic disease in hepatitis C infected populations Allison et al (1994) were the first to identify an interaction between chronic hepatitis C virus (HCV) infection and diabetes, demonstrating an increase in the prevalence of type 2 diabetes among HCV-infected patients with cirrhosis compared to patients with cirrhosis from other causes (50% versus 9%, respectively).1 Subsequent studies have found the prevalence of type 2 diabetes among this population to range between, 7.6% to 50%.2 The presence of insulin resistance and type 2 diabetes in HCV has been associated with poor HCV antiviral treatment response,3,4 acceleration of liver fibrosis,5 increased risk for hepatocellular carcinoma (HCC),6 higher transplant complication rates7 and possibly increased morbidity from cardiovascular and metabolic complications.8 Early intervention with lifestyle modification and/or metformin in patients with pre-diabetes can delay or prevent the onset of type 2 diabetes in high risk populations. It is unknown whether this benefit extends to those infected with HCV.9 [see Appendix I for definitions of insulin resistance, impaired fasting glucose, and diabetes] There is lack of agreement on how to manage insulin resistance in HCV-infected patients. There may be risks with some diabetes medications in this population. Sulfonylureas and insulin may be associated with an increased risk of developing HCC in this population. Additional evaluation of the risks and benefits of diabetic medications in HCV are required.10 HCV is also known to induce changes in lipid metabolism. The HCV life cycle is dependent on the VLDL pathway. Viral replication involves the formation of complexes termed lipoviral particles resulting in decreased secretion of VLDL. The assembly of these lipoviral particles is believed to facilitate binding with LDL receptor and considered a mechanism by which HCV gains entry to the hepatocyte. Numerous studies have demonstrated lower total cholesterol, triglycerides (TG), HDL-C and LDL-C levels in patients with chronic hepatitis C infection. Lower lipid levels correlate with higher HCV viral load,11 decreased antiviral virological cure rates12 [A.K.A Sustained Virological Response (SVR)] and increased hepatic steatosis.13,14 Successful treatment of HCV with IFN/Ribavirin is typically associated with the reversal of hypolipidemia yet in some patients lipid levels may increase to levels associated with increased cardiovascular risk.15,16

The metabolic effects of new HCV therapies are unknown in HCV-Infection Three HCV protease inhibitors (simeprevir, telaprevir, boceprevir) have been approved for the treatment of genotype 1 infection in combination with interferon and ribavirin. Telaprevir and simeprevir are dosed in combination with PEG-IFN and ribavirin for the initial 12 weeks of treatment. Interferon and ribavirin are dosed for 12 to 36 additional weeks based on early virological response and patient characteristics including liver fibrosis stage. Sofosbuvir is a nucleotide dosed in combination with pegylated interferon and ribavirin for 12 weeks in genotype 1 infected individuals. It can also be used in combination with simeprevir +/- ribavirin for 12 weeks without interferon. Sofosbuvir and ribavirin for 24 weeks is a third viable option of sofosbuvir-containing therapy in genotype 1 infection. Other orally administered HCV antivirals (protease inhibitors, nucleosides, non-nucleosides, assembly inhibitors) in development are effective against genotype 1 and other genotypes as well. Abbvie has developed a 12-week combination DAA regimen consisting of a HCV protease inhibitor (ABT-450 based with ritonavir), a NS5a inhibitor (ABT-267; Ombitasvir), a polymerase inhibitor (ABT-333; Dasabuvir) with or without ribavirin. This regimen was licensed in Canada in December 2014.

There are limited data evaluating the influence of HCV protease inhibitors, nucleotides and other direct acting antiviral (DAAs) drug classes on the metabolic milieu of HCV treatment recipients. In one study of HCV mono-infected study participants receiving 14 days of monotherapy with the protease inhibitor danoprevir, serum HCV RNA and HOMA-IR [Appendix I] correlated significantly (Spearman rho=0.379, p<0.0001).17 At baseline, mean serum HCV-RNA level and mean HOMA-IR score were 6.2±0.5 log10 IU/ml and 3.8±1.9, respectively. At the end of 14 days of Danoprevir monotherapy the mean decrease in HCV RNA was 2.2±1.3 log10 IU/ml (p<0.0001) in patients who received the active drug (n=40). Concurrent with this, the mean HOMA-IR score decreased by 1.6±1.1 (p<0.0001), with a close correlation between HOMA-IR improvement and viral load decline. In contrast, HCV-RNA and HOMA-IR remained unchanged in placebo recipients. The effect of HCV-protease inhibitors and other DAAs on glucose metabolism beyond 14 days of treatment has not been established.

With the development of DAA, the predictors of treatment response have evolved. However, phase 3 studies suggest that lower baseline LDL-C levels continue to be a predictor of treatment response to telaprevir triple therapy. The effect of interferon and ribavirin free regimens on lipid homeostasis has not been established and it is not known if baseline cholesterol levels remain a predictor of treatment outcomes with these regimens.

Why conduct this research? The above is compelling data supporting the pursuit of research into the effects of HCV antivirals on metabolic homeostasis. As a further rationale and justification, the experience with HIV antiretrovirals has clearly demonstrated that antiviral medications can produce profound changes in glucose metabolism, lipid profile and other measures of metabolic homeostasis. This establishes biological plausibility for this focus of research in HCV.

The new knowledge created from this research will:

1. Provide new information on the metabolic effects of the Abbvie 3D HCV antiviral regimen.
2. Provide insight as to whether there are metabolic advantages with RBV-free compared to RBV-containing HCV regimens. This is particularly relevant given the current uncertainty regarding the need for RBV in IFN-free, oral DAA regimens.
3. Provide insight into the impact of cirrhosis on metabolic milieu before, during and after HCV antiviral therapy

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA evidence of HCV infection
* Documented history of chronic HCV RNA infection with Genotype 1
* Able to provide informed consent
* Available for ongoing follow-up if required

Exclusion Criteria:

* <18 years old
* Evidence of decompensated liver disease
* HOMA IR< 2.0
* HIV seropositivity
* Chronic HBV/HIV infection
* Use of immune suppressing medications
* Active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Pilot Evaluation of the Influence of ABT450r, Ombitasvir, Dasabuvir +/- Ribavirin Hepatitis C Antiviral Therapy on Insulin Resistance | 30 weeks
  serial insulin sensitivity evaluation

SECONDARY OUTCOMES:
Pilot Evaluation of the Influence of ABT450r, Ombitasvir, Dasabuvir +/- Ribavirin Hepatitis C Antiviral Therapy Lipid Homeostasis | 30 weeks
  serial lipid homeostasis evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Publication Conference presentation Knowledge translation with community groups